CLINICAL TRIAL: NCT02066129
Title: Step-up Yellow Zone Inhaled Corticosteroids to Prevent Exacerbations
Acronym: STICS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, dave mauger, Principal Investigator, AsthmaNet Data Coordinating Center, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AsthmaNet 008
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: Asthma; Fluticasone
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluticasone 44 mcg (Active Comparator): Fluticasone 44 mcg 2 puffs twice daily for 7 days initiated at the onset of "yellow zone" symptoms.
  Interventions: Drug: Fluticasone 44 mcg
- Fluticasone 220 mcg (Active Comparator): Fluticasone 220 mcg 2 puffs twice daily for 7 days initiated at the onset of "yellow zone" symptoms.
  Interventions: Drug: Fluticasone 220 mcg

INTERVENTIONS:
Drug: Fluticasone 44 mcg — Fluticasone is an inhaled corticosteroid
  Other Names: Flovent® 44 mcg
  Arms: Fluticasone 44 mcg
Drug: Fluticasone 220 mcg — Fluticasone is an inhaled corticosteroid
  Other Names: Flovent® 220 mcg
  Arms: Fluticasone 220 mcg

SUMMARY:
The objective of this study is to determine whether, in children receiving low-dose inhaled corticosteroids (ICS), quintupling the dose of inhaled corticosteroids at the onset of symptoms previously associated with upper respiratory illnesses and subsequent asthma exacerbations reduces the rate of severe asthma exacerbations treated with oral corticosteroids.

DETAILED DESCRIPTION:
The study design is a double-blind, parallel-group trial, including a total of 250 participants, ages 5-11 years, with a diagnosis of asthma and a history of at least 1 asthma exacerbation treated with oral corticosteroids in the prior year. All participants will be treated for 48 weeks with open-label fluticasone 44 mcg 2 puffs twice daily. During the 48-week treatment period, participants will receive randomized blinded therapy for 7 days each time they enter the "yellow zone" (at the onset of symptoms previously associated with upper respiratory illnesses and subsequent asthma exacerbations). Yellow zone therapy will be fluticasone 44 or 220 mcg 2 puffs twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma
* At least 1 exacerbation treated with systemic (oral or injectable) corticosteroids in the past 12 months
* Able to perform reproducible spirometry
* Current treatment with step 2 controller therapy [low-dose ICS, leukotriene receptor antagonist (LTRA)] OR current treatment with step 3 controller therapy [low-dose ICS + long-acting beta agonist (LABA), low-dose ICS + LTRA, or medium dose ICS] with a childhood Asthma Control Test (c-ACT) score of >19, no more than 2 prednisone treated exacerbations in the past 6 months, prebronchodilator Forced Expiratory Volume at 1 second (FEV1) ≥ 80% predicted and willing to step down therapy OR controller naïve and qualifying for step 2 controller therapy [asthma symptoms or short acting beta agonist (SABA) use > 2 days per week or night-time awakenings due to asthma > 2 nights per month]
* Prebronchodilator FEV1 ≥ 60% predicted
* Ability and willingness to provide informed assent
* For females of childbearing potential: not pregnant, non-lactating, and agree to practice an adequate birth control method.
* History of clinical varicella or varicella vaccine

Exclusion Criteria:

* Systemic (oral or injectable) corticosteroids within previous 2-week period
* Current or recent (previous 2-weeks) use of medications known to significantly interact with corticosteroid disposition, including but not limited to carbamazepine, erythromycin, phenobarbital, phenytoin, rifampin, and ketoconazole
* Presence of chronic or active lung disease other than asthma
* Significant medical illness other than asthma, including thyroid disease, diabetes mellitus, Cushing's disease, Addison's disease, hepatic disease, or concurrent medical problems that could require oral corticosteroids during the study
* A history of cataracts, glaucoma, or any other medical disorder associated with an adverse effect to corticosteroids
* History of a life-threatening asthma exacerbation requiring intubation, mechanical ventilation, or resulting in a hypoxic seizure
* More than 5 prednisone treated exacerbations in the past 12 months
* More than 1 hospitalizations lasting >24 hours for asthma in the past 12 months
* History of adverse reactions to ICS preparations or any of their ingredients
* Receiving hyposensitization therapy other than an established maintenance regimen (On maintenance regimen for ≥ 3 months)
* History of premature birth before 35 weeks gestation

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 254 (Actual)
Dates: Start 2014-07; Primary Completion 2017-04-21 (Actual); Study Completion 2017-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Busse, MD, Study Chair — University of Wisconsin, Madison
Locations (18):
- United States (18):
  - University of Arizona College of Medicine, Tucson, Arizona
  - Children's Hospital & Research Center Oakland, Oakland, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center/Stroger Hospital, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Ann and Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Rainbow Babies and Children's Hospital, Case Western Reserve University, Cleveland, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Gomez LF, Kinnee E, Kaufman JD, Young MT, Fitzpatrick AM, Phipatanakul W, Mauger DT, McClure LA, Bilal U, Holguin F, Clougherty JE. Modification of asthma treatment efficacy by healthcare access: A reanalysis of AsthmaNet Step-Up Yellow Zone Inhaled Corticosteroids to Prevent Exacerbations (STICS) clinical trial. Respir Med. 2024 Nov-Dec;234:107853. doi: 10.1016/j.rmed.2024.107853. Epub 2024 Nov 5. PMID 39510322
- [Derived] Yuan H, Liu Z, Dong J, Bacharier LB, Jackson D, Mauger D, Boushey H, Castro M, Durack J, Huang YJ, Lemanske RF Jr, Storch GA, Weinstock GM, Wylie K, Covar R, Fitzpatrick AM, Phipatanakul W, Robison RG, Beigelman A, Zhou Y. The Fungal Microbiome of the Upper Airway Is Associated With Future Loss of Asthma Control and Exacerbation Among Children With Asthma. Chest. 2023 Aug;164(2):302-313. doi: 10.1016/j.chest.2023.03.034. Epub 2023 Mar 30. PMID 37003356
- [Derived] Jackson DJ, Bacharier LB, Mauger DT, Boehmer S, Beigelman A, Chmiel JF, Fitzpatrick AM, Gaffin JM, Morgan WJ, Peters SP, Phipatanakul W, Sheehan WJ, Cabana MD, Holguin F, Martinez FD, Pongracic JA, Baxi SN, Benson M, Blake K, Covar R, Gentile DA, Israel E, Krishnan JA, Kumar HV, Lang JE, Lazarus SC, Lima JJ, Long D, Ly N, Marbin J, Moy JN, Myers RE, Olin JT, Raissy HH, Robison RG, Ross K, Sorkness CA, Lemanske RF Jr; National Heart, Lung, and Blood Institute AsthmaNet. Quintupling Inhaled Glucocorticoids to Prevent Childhood Asthma Exacerbations. N Engl J Med. 2018 Mar 8;378(10):891-901. doi: 10.1056/NEJMoa1710988. Epub 2018 Mar 3. PMID 29504498
- See also: AsthmaNet — http://asthmanetresearch.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluticasone 44 mcg | Fluticasone 220 mcg
Started | 127 | 127
Completed | 98 | 94
Not Completed | 29 | 33
Not completed — Lost to Follow-up | 13 | 12
Not completed — Withdrawal by Subject | 7 | 10
Not completed — Lack of Efficacy | 8 | 10
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone 44 mcg | Fluticasone 220 mcg | Total
Number analyzed (Participants) | 127 | 127 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (1.9) | 8.1 (1.8) | 8.0 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 44 | 91
  Male | 80 | 83 | 163
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 64 | 76 | 140
  Black | 29 | 27 | 56
  Other | 34 | 24 | 58
Region of Enrollment [Number; unit: participants]
  United States | 127 | 127 | 254
Blood eosinophils [Mean (Standard Deviation); unit: cells per cubic millimeter] | 367 (300) | 327 (234) | 346 (268)
Number of positive allergen specific IgE tests [Mean (Standard Deviation); unit: count] | 4.8 (4.2) | 5.2 (4.5) | 5.0 (4.4)
Hospitalized in year prior to enrollment [Count of Participants; unit: Participants] | 16 | 15 | 31
Post albuterol forced expiratory volume at one second (FEV1) % of predicted [Mean (Standard Deviation); unit: percent] — FEV1 following 4 puffs of albuterol, expressed as percent of predicted (based on age, sex, race, and height).
  percent | 106.8 (15.6) | 107.8 (13.9) | 107.3 (14.8)
At least one allergen specific immunoglobulin E (IgE) tests [Count of Participants; unit: Participants] | 88 | 99 | 187

OUTCOME MEASURES:

1. Primary Outcome: Asthma Exacerbations
Description: The primary outcome is the rate of severe asthma exacerbations treated with oral corticosteroids during the 48 week treatment period.
Time Frame: end of 48 week treatment period
Measure: Least Squares Mean (95% Confidence Interval); unit: exacerbations per year
Arm/Group | Fluticasone 44 mcg | Fluticasone 220 mcg
Number analyzed (Participants) | 127 | 127
exacerbations per year | 0.37 [0.25 to 0.55] | 0.48 [0.33 to 0.70]

2. Secondary Outcome: Yellow Zone Asthma Symptoms
Description: Study participants completed a daily symptom diary. They scored the following diary elements on a scale from 0-3 (none-severe): Cough, Wheeze, Trouble Breathing, Interference With Activities. A combined score was calculated as the sum of the 4 elements and ranged from 0 to 12. The study intervention was based on yellow-zones as noted in the Study Description. This outcome was based on diary data including 21 days, beginning 7 days prior to the onset of the yellow-zone intervention and ending 14 days after the onset of the intervention. The total symptom burden outcome was defined as the sum of the combined score on each diary day and ranged from 0 to 252 (max combined score of 12 per day multiplied by 21 days). A score of zero would indicate no symptoms over the entire 21 days. A score of 252 would indicate severe cough, wheeze, shortness of breath, and interference with activities on all of the 21 days.
Time Frame: end of 48 week treatment period
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fluticasone 44 mcg | Fluticasone 220 mcg
Number analyzed (Participants) | 127 | 127
units on a scale | 20 [17 to 24] | 23 [19 to 27]

3. Secondary Outcome: Yellow Zone Albuterol Use
Description: Use of albuterol rescue medication during 7-day yellow zone episodes.
Time Frame: end of 48 week treatment period
Measure: Least Squares Mean (95% Confidence Interval); unit: number of albuterol puffs
Arm/Group | Fluticasone 44 mcg | Fluticasone 220 mcg
Number analyzed (Participants) | 127 | 127
number of albuterol puffs | 13 [11 to 16] | 15 [13 to 19]

4. Secondary Outcome: Unscheduled Emergency Department (ED) or Urgent Care Visits for Asthma
Description: Rate of emergency department (ED) or urgent care visits for asthma during the 48 week treatment period.
Time Frame: end of 48 week treatment period
Measure: Least Squares Mean (95% Confidence Interval); unit: visits per year
Arm/Group | Fluticasone 44 mcg | Fluticasone 220 mcg
Number analyzed (Participants) | 127 | 127
visits per year | 0.47 [0.31 to 0.72] | 0.64 [0.42 to 0.96]

5. Secondary Outcome: Number of Participants Hospitalized for Asthma
Description: Number of participants hospitalized for asthma during the 48 week treatment period.
Time Frame: end of 48 week treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Fluticasone 44 mcg | Fluticasone 220 mcg
Number analyzed (Participants) | 127 | 127
Participants | 0 | 4

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Fluticasone 44 mcg | Fluticasone 220 mcg
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/127
Serious Adverse Events (participants affected / at risk) | 1/127 | 4/127
Other Adverse Events (participants affected / at risk) | 115/127 | 111/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluticasone 44 mcg (N=127) | Fluticasone 220 mcg (N=127)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Hypertrophy Tonsils/Adenoids (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluticasone 44 mcg (N=127) | Fluticasone 220 mcg (N=127)
Otitis media (Nervous system disorders) | 14 (17) | 14 (20)
Acute nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 46 (99) | 33 (57)
Acute respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 22 (39) | 21 (41)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 7 (9)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 36 (62) | 28 (45)
Infectious enteritis (Infections and infestations) | 7 (8) | 6 (7)
Strep sore throat (Infections and infestations) | 5 (5) | 10 (16)
Cough (General disorders) | 29 (45) | 30 (49)
Fever (General disorders) | 24 (39) | 21 (28)
Headache (General disorders) | 15 (22) | 10 (12)
Throat pain (General disorders) | 5 (7) | 8 (8)
Vomiting alone (General disorders) | 8 (9) | 10 (14)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 6 (8)
Acute asthma attack (Respiratory, thoracic and mediastinal disorders) | 25 (32) | 30 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT02066129/Prot_SAP_000.pdf